CLINICAL TRIAL: NCT03765814
Title: Paramedical Evaluation of a Standardize Procedure of Selection of Serious Brain-injured Patients in Therapeutic Abstention to a Brain Death State in the First 48h
Brief Title: The Anticipated Organ Donation Approach
Acronym: PREMORENCE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-CHITS-02; 2018-A01455-50 (Other: Id-RCB)
Record Dates: First submitted 2018-11-22; First posted 2018-12-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Brain Death
Keywords: organ donation; serious brain-injured patient; anticipated approach
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to make a paramedical evaluation of a selection procedure of serious brain-injured patient in therapeutic abstention to a brain death state within 48 hours.

DETAILED DESCRIPTION:
In 2016 in France, 5891 organs have been transplanted. All the transplant's sources are developed (brain death, Maastricht III, living organ donor).

However, the French Transplant's plan 2017-2021 require always more transplant, the aim is to reach 7800 transplants in 4 years.

To increase the number of transplants, one of the strategies is to actively identify the donors in brain death state and the donors with wider criteria. It's mainly serious brain-injured patients.

The procedure of early announcement of organ donation consists in beginning or pursues intensive care on serious brain-injured patient, for whom a decision of abstention of therapeutic active was decided. The only purpose of the medical care is to notice the brain death state that lead to donation.

In 2010, an expert group of the "Société de reanimation de langue Française" established guidelines to manage organ's donation in serious brain-injured patient after a stroke. The interest, to admit these serious brain-injured patients in intensive care unit, is to increase the number of donors in state of brain death and so the number of transplants.

However the guidelines remain little practised and little known in France. The number of bed in intensive care unit is limited and requires a selection of the potential organ donors. To hospitalised serious brain-injured patients in intensive care unit, there are no validated selection criteria that make difficult the implication of the transplant coordination in this anticipated announcement's approach.

In Toulon hospital, a standardize selection procedure was initiated and applied systematically by the transplant coordinator for each serious brain-injured patients. The selected patients will evolve in brain death state in 48 hours and could be organ donors.

The aim of this study is to validate a paramedical procedure to increase the number of organ donors.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female over 18 years-old
* Patient with serious brain damages
* Medical decision of withdrawing life sustaining treatment
* Signed and dated informed consent by trusted person, or family
* Patient covered by social security regimen
* Patient eligible for organ donation according to organ donation hospital co-ordination
* Glasgow Coma Scale (GCS) :

  * Seriously brain-injured patient without confounding factors, head trauma, brain anoxia or ischemic stroke : GCS<5 and loss of bilateral corneal reflex or GCS<5 and loss of three brain stem reflexes
  * Seriously brain-injured patient with confounding factors and without head trauma, brain anoxia or ischemic stroke : at least one of the following scanographic sign of gravity : deletion of subarachnoid cisterns, more than 15 mm deviation of the median line, hematoma volume > 65 cm3 or hydrocephalus due to intra-ventricular bleeding with V3 or V4 flood, and, if documented, a GCS<7.
  * Patient with head trauma, brain anoxia or ischemic stroke, reliable clinical examination required (no confounding factor) : GCS<5 and loss of bilateral corneal reflex or GCS<5 and loss of three brain stem reflexes

Exclusion Criteria:

* No trusted person or family present
* Seriously brain-injured patient because of head trauma, brain anoxia or ischemic stroke with confounding factors
* Absolute contraindication to organ donation known at the moment of inclusion (HIV, rabies, active cancer, active tuberculosis, Creutzfeldt-Jakob disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Seriously brain-injured patient with therapeutic abstention
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2019-09-29 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Study of the evolution to brain death state within 48 hours of seriously brain-injured patients selected by a standardized procedure and hospitalised in intensive care unit. | 48 hours after validation of eligibility
  Rate of patients evolving to brain death state during the first 48 hours following the examination which validates patient's eligibility

SECONDARY OUTCOMES:
Evaluation of call rate to transplant coordination that don't result in a procedure of anticipated announcement | 48 hours after validation of eligibility
  Ratio between the number of non-eligible patients and the total number of calls
Evaluation of close family refusal rate for pursuit of care during 48h in intensive care unit | 48 hours after validation of eligibility
  Ratio between the number of family refusal and the total number of patients for whom the anticipated announcement procedure was started.
Number of refusal causes in the population | 48 hours after validation of eligibility
  Number of refusal causes will be presented globally
Evaluation of the delay between eligibility validation and the passage in brain death state. | 48 hours after validation of eligibility
  The passage delay between eligibility validation and brain death state is defined by the time in hours between the examination which validates patient's eligibility and the diagnosis of brain death state.
Evaluation of the rate of patients with organ removal in enrolled patients. | 48 hours after validation of eligibility
  Ratio between the number of patient who performed organ donation and the total number of patients included.
Number and type of organ harvested by patient. | 48 hours after validation of eligibility
  Number of organs collected will be presented globally, by patient and by type of organ transplanted.
Number of transplants performed. | 10 days
  The number of transplants performed will be presented globally, by patient and by type of organs.
Number of patient enrolled by type of service. | 48 hours after validation of eligibility
  The number of patient enrolled in the intensive care unit, the Emergency or Neurovascular intensive care unit will be described globally
Non harvested organs which have been suggested for transplant | 10 days
  The proportion of suggested non harvested organs will be determined as the number of suggested non harvested organs divided by the total number of non harvested organs. Reasons of suggested organs refusal will be presented.
Number of patients who performed Maastricht 3 organ donation among patients who didn't evolve to brain death state | 10 days
  The rate of patients with Maastricht 3 organ donation will be determined as the number of patients having performed Maastricht 3 organ donation divided by the number of patients who didn't evolve to brain death state after 48hours

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Arsonneau, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (4):
- France (4):
  - CH Annecy Genevois, Pringy, Haute Savoie
  - CHU de Nantes, Nantes, Loire-Atlantique
  - Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, Toulon, Var
  - Centre Hospitalier Départemental de Vendée Les Oudairies, La Roche-sur-Yon, Vendée

IPD SHARING:
Plan to Share IPD: No
no plan